CLINICAL TRIAL: NCT03164161
Title: The Relationship Between Saliva β-endorphins Levels, Sensitivity and Tolerance to Cold Pain and Perception of Pain in Oral Surgery Procedures in Adult Patients
Brief Title: The Relationship Between Saliva β-endorphins Levels, Cold Pressor Test and Perception of Pain in Oral Surgery Procedures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Lithuanian University of Health Sciences (Other)
Responsible Party: Principal Investigator, Inesa Astramskaitė, Principal investigator, Lithuanian University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: BEC-OF-8
Record Dates: First submitted 2016-09-29; First posted 2017-05-23 (Actual); Last update posted 2017-05-23 (Actual); Status verified 2017-05

CONDITIONS: Hyperalgesia; Pain Insensitivity, Congenital
Keywords: Pain Sensitivity; Measurement; Cold Pressor; β-endorphins; saliva; oral surgery
MeSH Terms: conditions — Hyperalgesia; Pain Insensitivity, Congenital

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cold Pressor Test Results (Active Comparator): Participants, enrolling the healthy participants high and low pain perception groups, will undergo cold pressor test. According to the results patients will be assigned according to time (min:s) until first pain felt (pain threshold) and time (min:s) until unbearable pain and test withdraw (pain tolerance). Also, pain ratings (1-10) at same points will be used as participants alignment tool.
  Interventions: Device: Cold pressor test
- β-endorphins level in saliva (Active Comparator): Participants will be sorted according to β-endorphin levels in saliva., therefore the β-endorphins evaluation in saliva intervention will be performed.
  Interventions: Other: β-endorphins evaluation in saliva
- β-endorphin level in blood plasma (Active Comparator): Participants will be sorted according to β-endorphin levels in blood plasma, therefore β-endorphins evaluation in blood plasma will be performed.
  Interventions: Other: β-endorphins evaluation in blood plasma
- Pain perception rating (No Intervention): Healthy participants will be sorted in to groups: high and low pain perception groups, according to the results of questionnaires, containing various oral surgery procedures pain ranking.

INTERVENTIONS:
Device: Cold pressor test — Described before.
  Arms: Cold Pressor Test Results
Other: β-endorphins evaluation in saliva — Described before.
  Arms: β-endorphins level in saliva
Other: β-endorphins evaluation in blood plasma — Described before.
  Arms: β-endorphin level in blood plasma

SUMMARY:
The purpose of this study is to evaluate the correlation between β-endorphin levels in blood plasma and saliva in healthy participants with different pain sensitivity and in those with acute pain in oral and maxillofacial region.

Expected results

* Relation between blood plasma and saliva β-endorphins levels
* Differences of blood plasma β-endorphins levels in healthy participants with different pain sensitivity and in those with acute pain
* Differences of saliva β-endorphins levels in healthy participants with different pain sensitivity and in those with acute pain
* Objective method of patient's pain sensation evaluation
* Correlation between patient's self-reported understanding of pain levels in oral surgery procedures, levels in saliva and blood plasma β-endorphins levels and sensitivity to cold test results

Study protocol:

Selection of participants

1. Evaluation of pain perception in oral surgery procedures by healthy adult participants.
2. Groups formation, according to the results from first stage, resulting in high and low pain rating participants groups.
3. Control group formation from patients with acute pain in oral and maxillofacial region Control rating of participants

1. Patients that have been assigned to groups according to subjective pain ratings in oral surgery procedures will have to repeat the same questionnaire to ensure the correct group assignment.

2. Patients that have been assigned to groups according to subjective pain ratings in oral surgery procedures, will undergo the sensitivity and tolerance to cold pain test.

3. Patients that were assigned to control-acute pain group, will be included in further study stages only with clinically diagnosed cause of acute pain in oral and maxillofacial region to avoid possible psychogenic or general diseases pain.

Evaluation of β-endorphins - sampling

1. Saliva samples will be collected by all further included participants by one selves participants with researchers supervision.
2. Blood samples will be collected from forearm veins by researcher. Evaluation of β-endorphins - laboratorial examination

1. Levels of β-endorphins in saliva and blood will be evaluated according to manufacturer of β-endorphins evaluation kit for human research. Every sample will be evaluated twice and the mean level will be evaluated.

Statistical analysis

1. Statistical analysis will be produced to access all possible relationships

DETAILED DESCRIPTION:
Fear of dental pain, despite the modern analgesia methods, is still a trigger for many patients, resulting in fear of dentistry. Pain and anxiety during the oral surgery procedures are related to each other. Since fear is a multi-caused state, it is important to analyse each causing factor. Pain sensitivity, or fear of pain, in dental office is different in each person because of various psychological aspects, but also because of genetic code. Pain mechanism is a complex system with many different pathways, resulting in possibility to feel pain. It is interesting that despite the anxiety and stress having a positive correlation with perceived pain, high stress levels may reduce the pain sensation. Stress mechanism involves pain regulation, which may result in hyperalgesia or analgesia. During the stress many organ systems are activated, including the hypothalamic secretion of beta-endorphins, causing analgesia. Therefore, beta-endorphins are secreted by pituitary gland and then spreads to all body by diffusion. However, some studies suggest that beta-endorphins can be also produced by immune cells during the inflammation. Beta-endorphins act like natural morphines, binding the mu-receptors and activating the pain reduction system, therefore beta-endorphin plasma levels correlates with expressed pain. Various studies suggest that low level of peripheral plasma beta-endorphin levels act in chronic pain and trigeminal neuralgia development. Beta-endorphins have also been found as predictive factors to set the overtraining in sports, which result in muscles overloading because of euphoric and analgesic effects. Therefore, investigators have hypothesised that beta-endorphins could be a reliable factor determining patient's pain sensitivity or chronical non-painful processes. Also, since pain rating is usually based on self-reported questionnaires, beta-endorphins evaluation may be possible objective pain evaluation. However, most studies evaluating beta-endorphins levels are based on blood samples evaluation, and blood sampling is a painful and stressful event by itself. Beta-endorphins can also be assessed in saliva, however no previous studies have evaluated the relation between saliva beta-endorphins and plasma beta-endorphins in patients with different pain sensitivity. The aim of this study is to evaluate the relationship between plasma beta-endorphin and saliva beta-endorphin levels in patients with different pain sensitivity and patients with acute pain in maxillofacial region.

Study design

* Assessment: Healthy participants will be assessed in two groups regarding the evaluation of pain in common procedures in oral surgery self-reported questionnaire. The questionnaire is composed from 10 items, including perception of pain during surgical procedures and perception of post-operative healing caused pain. Procedures, such as anaesthetic injection, wisdom tooth removal, mobile tooth extraction, stitches removal, implantation and incision are composed into questionnaire. All items must be rated in numerical rating scales (NRS) from 1 - no pain to 10 - extreme pain, according to patient's assumption. Participants to further clinical trial will be randomly selected to form two groups with low and high pain rating. Further involved participants will have to repeat pain rating questionnaires to avoid possible accidental items rating. Cold pressor test will be enrolled for both groups in further described method.
* Cold pressor test. Participants will have to hold their hand up to the wrist in 5° temperature water, since it was suggested as a medium temperature giving the results of appropriate test time and felt pain. The water temperature below 15°C is known to stimulate nociceptors and provoke pain, however the testing time is relatively to long and the minimum temperature to this test of -2°C quickly provokes pain and it encumbers time evaluation. Digital thermometer will be used to ensure even temperature during the test with error of 0,5°C. The time of first painful sensation (pain threshold) will be noted and patients will be asked to self-report the felt pain in 1-10 NRS, afterwards the time of hand withdraw will be also recorded (pain tolerance) and the pain will be rated as described before. The maximum time of the test will be 4 minutes. If at the end of 4 minutes patient is still continuing, he will be asked to rate pain felt at 4 minutes moment in 10 points NRS and the test will be withdraw.
* Patients to control - acute pain group will be assessed randomly from those, coming for help because of acute pain in oral and maxillofacial region. Patients will be asked to voluntarily participate in research, with the aim of best patient's care and least interference to the needed treatment procedures. Only patients with clinically diagnosed cause of acute pain will be enrolled, even though it is stated that pain is present for patient, whenever a patient reports pain, with the aim to avoid any psychogenic pain. Also, patients will be asked to rate their present pain in NRS and only those assessing pain not less than 4 out of 10 points will be further included, since it is described as moderate pain at 4-6 points and severe pain at 7-10 points. Also, NRS is known as appropriate numerical method, if pain is empirically tested.
* Β-endorphins evaluation. Participants from non-acute-pain group will be tested the other day than cold-pressor test to eliminate the effect of pain pressor test stimulated stress, resulting in sympathetic system activation, including β-endorphins production. Before the sampling patients will be asked to calm and stay still until they feel relaxed to avoid possible stress effect on results. The saliva samples will be collected by participants with researcher's supervision in sterile test-tubes. It is known that β-endorphins can be found in saliva, however it is not commonly used in pain evaluating researches. Afterwards the blood sampling will be provided with the aim not to produce blood collection caused stress before saliva sampling. Blood samples will be used as control samples to ensure the presence of β-endorphins in organism at exact moment and to rate the blood β-endorphins concentrations relation with saliva β-endorphin levels.
* Β-endorphins sampling in control - acute pain group will be provided at the same day as acute pain is felt. This group will be used as control, since it is presumed that acute pain and stress increases β-endorphins levels. Saliva sample will be collected by participant under the researcher's supervision. Afterwards the blood sample will be collected.
* Laboratorial examination. Will be performed according to manufacturer's recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Patients without reported chronical or acute pain in non-acute-pain group
* Patients with acute pain in oral and maxillofacial region with diagnosed cause of pain in acute-pain group
* Patients older than 18 years

Exclusion Criteria:

* Patients undertaking any pain relieving medicine, including non-steroid and opioid medicine
* Patients with diagnosed endocrine system diseases
* Patients with psychogenic diseases
* Patients with pre-injected local anaesthetics
* Patients with oncologic diseases
* Patients with endocrine system diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-05 (Estimated); Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Correlations between β-endorphins levels (pg/mL) and cold pressor test (min:s), pain perception (1-10 points) questionnaire results. | One year
  Both, saliva and blood β-endorphins levels will be compared with cold pressor test results and pain perception in oral surgery test results. Blood β-endorphin levels will be used only as control measurement, focusing on saliva β-endorphin levels correlation.

SECONDARY OUTCOMES:
Differences between acute-pain group and healthy participants groups with different pain sensitivity levels | One year
  All data will be compared between acute-pain and healthy participants groups, to determine, if acute-pain causes β-endorphin levels change.
Correlation between saliva β-endorphins and blood plasma β-endorphins levels | One day
  Correlations between saliva and blood plasma β-endorphin levels will be calculated with the necessity to collect both samples at the same day and to do laboratorial examinations twice for each sample.
Correlation between pain perception in oral surgery questionnaire and cold pressor test results | One year
  Possible correlations between pain perception in oral surgery questionnaire results and various results from cold pressor test will be calculated. Time (min:s) and pain rating points (1-10) will be taken from cold pressor test and compared with questionnaires points sum (1-100)
Pain perception in oral surgery questionnaire test - retest correlation | One year
  Correlation between primary questionnaire rating and secondary questionnaire rating on pain pressor test day will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Gintaras Juodžbalys, PhD, Study Chair — Lithuanian Universwity of Health Sciences; Rasa Banienė, Study Chair — Lithuanian University of Health Sciences

IPD SHARING:
Plan to Share IPD: No
No individual data will be available for sharing.

REFERENCES:
- [Background] Sanikop S, Agrawal P, Patil S. Relationship between dental anxiety and pain perception during scaling. J Oral Sci. 2011 Sep;53(3):341-8. doi: 10.2334/josnusd.53.341. PMID 21959662
- [Background] Kyle BN, McNeil DW, Weaver B, Wilson T. Recall of Dental Pain and Anxiety in a Cohort of Oral Surgery Patients. J Dent Res. 2016 Jun;95(6):629-34. doi: 10.1177/0022034516631977. Epub 2016 Feb 23. PMID 26908629
- [Background] Randall CL, McNeil DW, Shaffer JR, Crout RJ, Weyant RJ, Marazita ML. Fear of Pain Mediates the Association between MC1R Genotype and Dental Fear. J Dent Res. 2016 Sep;95(10):1132-7. doi: 10.1177/0022034516661151. PMID 27555332
- [Background] Klages U, Ulusoy O, Kianifard S, Wehrbein H. Dental trait anxiety and pain sensitivity as predictors of expected and experienced pain in stressful dental procedures. Eur J Oral Sci. 2004 Dec;112(6):477-83. doi: 10.1111/j.1600-0722.2004.00167.x. PMID 15560829
- [Background] Astramskaite I, Poskevicius L, Juodzbalys G. Factors determining tooth extraction anxiety and fear in adult dental patients: a systematic review. Int J Oral Maxillofac Surg. 2016 Dec;45(12):1630-1643. doi: 10.1016/j.ijom.2016.06.019. Epub 2016 Jul 18. PMID 27436789
- [Background] Duan G, Han C, Wang Q, Guo S, Zhang Y, Ying Y, Huang P, Zhang L, Macala L, Shah P, Zhang M, Li N, Dib-Hajj SD, Waxman SG, Zhang X. A SCN10A SNP biases human pain sensitivity. Mol Pain. 2016 Sep 2;12:1744806916666083. doi: 10.1177/1744806916666083. Print 2016. PMID 27590072
- [Background] Basbaum AI, Bautista DM, Scherrer G, Julius D. Cellular and molecular mechanisms of pain. Cell. 2009 Oct 16;139(2):267-84. doi: 10.1016/j.cell.2009.09.028. PMID 19837031
- [Background] National Research Council (US) Committee on Recognition and Alleviation of Pain in Laboratory Animals. Recognition and Alleviation of Pain in Laboratory Animals. Washington (DC): National Academies Press (US); 2009. Available from http://www.ncbi.nlm.nih.gov/books/NBK32658/ PMID 20662126
- [Background] Amit Z, Galina ZH. Stress-induced analgesia: adaptive pain suppression. Physiol Rev. 1986 Oct;66(4):1091-120. doi: 10.1152/physrev.1986.66.4.1091. PMID 2876446
- [Background] Ahmad AH, Zakaria R. Pain in Times of Stress. Malays J Med Sci. 2015 Dec;22(Spec Issue):52-61. PMID 27006638
- [Background] Dalayeun JF, Nores JM, Bergal S. Physiology of beta-endorphins. A close-up view and a review of the literature. Biomed Pharmacother. 1993;47(8):311-20. doi: 10.1016/0753-3322(93)90080-5. PMID 7520295
- [Background] Sprouse-Blum AS, Smith G, Sugai D, Parsa FD. Understanding endorphins and their importance in pain management. Hawaii Med J. 2010 Mar;69(3):70-1. No abstract available. PMID 20397507
- [Background] Backryd E, Ghafouri B, Larsson B, Gerdle B. Do low levels of beta-endorphin in the cerebrospinal fluid indicate defective top-down inhibition in patients with chronic neuropathic pain? A cross-sectional, comparative study. Pain Med. 2014 Jan;15(1):111-9. doi: 10.1111/pme.12248. Epub 2013 Oct 4. PMID 24118997
- [Background] Zhao YF, Jiang XZ, Hu SH, Liu Y, Miao L, Song CY. [Observation of plasma levels of beta-endorphin in patients with trigeminal neuralgia]. Shanghai Kou Qiang Yi Xue. 2001 Mar;10(1):46-8. Chinese. PMID 14994078
- [Background] Cunha GS, Ribeiro JL, Oliveira AR. [Levels of beta-endorphin in response to exercise and overtraining]. Arq Bras Endocrinol Metabol. 2008 Jun;52(4):589-98. doi: 10.1590/s0004-27302008000400004. Portuguese. PMID 18604371
- [Background] Saltychev M, Vastamaki H, Mattie R, McCormick Z, Vastamaki M, Laimi K. Psychometric Properties of the Pain Numeric Rating Scale When Applied to Multiple Body Regions among Professional Musicians. PLoS One. 2016 Sep 7;11(9):e0161874. doi: 10.1371/journal.pone.0161874. eCollection 2016. PMID 27603011
- [Background] Gill HS, Prausnitz MR. Does needle size matter? J Diabetes Sci Technol. 2007 Sep;1(5):725-9. doi: 10.1177/193229680700100517. PMID 19885141
- [Background] Rai B, Kaur J. Salivary stress markers and psychological stress in simulated microgravity: 21 days in 6 degrees head-down tilt. J Oral Sci. 2011 Mar;53(1):103-7. doi: 10.2334/josnusd.53.103. PMID 21467821
- [Background] Wolf S, Hardy JD. STUDIES ON PAIN. OBSERVATIONS ON PAIN DUE TO LOCAL COOLING AND ON FACTORS INVOLVED IN THE "COLD PRESSOR" EFFECT. J Clin Invest. 1941 Sep;20(5):521-33. doi: 10.1172/JCI101245. No abstract available. PMID 16694857
- [Background] Mitchell LA, MacDonald RA, Brodie EE. Temperature and the cold pressor test. J Pain. 2004 May;5(4):233-7. doi: 10.1016/j.jpain.2004.03.004. PMID 15162346
- [Background] Koenig J, Jarczok MN, Ellis RJ, Bach C, Thayer JF, Hillecke TK. Two-week test-retest stability of the cold pressor task procedure at two different temperatures as a measure of pain threshold and tolerance. Pain Pract. 2014 Mar;14(3):E126-35. doi: 10.1111/papr.12142. Epub 2013 Nov 20. PMID 24256148
- [Background] Lovallo W. The cold pressor test and autonomic function: a review and integration. Psychophysiology. 1975 May;12(3):268-82. doi: 10.1111/j.1469-8986.1975.tb01289.x. No abstract available. PMID 1153632
- [Background] V Nikolov, M Petkova, B Petrova, K Mineva. Pain perception to the cold pressor test in reproductive - age women: relation to menstrual phase and comparison with men. Trakia J Sci. 12(1):376-380, 2014
- [Background] Herr K, Coyne PJ, McCaffery M, Manworren R, Merkel S. Pain assessment in the patient unable to self-report: position statement with clinical practice recommendations. Pain Manag Nurs. 2011 Dec;12(4):230-50. doi: 10.1016/j.pmn.2011.10.002. PMID 22117755
- [Background] Pain: clinical manual for nursing practice Pain: clinical manual for nursing practice Margo McCaffery Alexander Beebe Mosby Yearbook UK pound17.25 0 7234 1992 2. Nurs Stand. 1994 Dec 7;9(11):55. doi: 10.7748/ns.9.11.55.s69. PMID 27527475
- [Background] Hjermstad MJ, Fayers PM, Haugen DF, Caraceni A, Hanks GW, Loge JH, Fainsinger R, Aass N, Kaasa S; European Palliative Care Research Collaborative (EPCRC). Studies comparing Numerical Rating Scales, Verbal Rating Scales, and Visual Analogue Scales for assessment of pain intensity in adults: a systematic literature review. J Pain Symptom Manage. 2011 Jun;41(6):1073-93. doi: 10.1016/j.jpainsymman.2010.08.016. PMID 21621130
- [Background] Mourot L, Bouhaddi M, Regnard J. Effects of the cold pressor test on cardiac autonomic control in normal subjects. Physiol Res. 2009;58(1):83-91. doi: 10.33549/physiolres.931360. Epub 2008 Jan 17. PMID 18198985